CLINICAL TRIAL: NCT07346365
Title: Spontaneous Dislocation and Adverse Events of a Prophylactic Pancreatic Stent: a Prospective, Randomised, Multicenter Study (SAFE PANCREAS)
Brief Title: Spontaneous Dislocation and Adverse Events of a Prophylactic Pancreatic Stent
Acronym: SAFE PANCREAS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: SRH Wald-Klinikum Gera GmbH (Other); Asklepios Kliniken Hamburg GmbH (Other); Charité - Universitätsmedizin Berlin, Campus Virchow Klinikum (Unknown); Helios Klinikum Krefeld (Unknown); Sana Klinikum Offenbach (Other); St. Josef Hospital Bochum (Other); University Hospital, Aachen (Other); University Hospital, Essen (Other); University Hospital Freiburg (Other); Münster University Hospital, Germany (Unknown); Medizinische Universitätsklinik Tübingen (Unknown); University of Göttingen (Other); University Hospital, Basel, Switzerland (Other); Centrum Gastroenterologie Bethanien (Unknown); University Hospital Munich (LMU) (Unknown); Universitätsklinik Würzburg (Unknown)
Responsible Party: Principal Investigator, Georg Dultz, Senior Physician at Clinic of Gastroenterology, Johann Wolfgang Goethe University Hospital, Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FloMi2025
Record Dates: First submitted 2025-11-25; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Stent Dislodgement; ERCP; Pancreas Stent; Post-ERCP Pancreatitis; Prophylactic Pancreatic Stent
Keywords: ercp; prophylactic pancreatic stent; post-ercp-pancreatitis; pancreatic stent; post-ercp pancreatitis; PEP

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (Active Comparator): Standard time of the removal
  Interventions: Device: standard group
- Interventional - delayed removal (Experimental): Stent removal after 1 - 3 months
  Interventions: Device: pancreatic stent removal

INTERVENTIONS:
Device: pancreatic stent removal — Removal of the pancreatic stent after 1 - 3 months after the placement
  Arms: Interventional - delayed removal
Device: standard group — Removal at intervals of 12 hours up to a maximum of 10 days after the index ERCP
  Arms: Standard

SUMMARY:
A multicenter, prospective, controlled randomized study to investigate the optimal duration of protective pancreatic stents after endoscopic retrograde cholangiopancreatography (ERCP).

The primary endpoint is the complication rate that can be clinically attributed to the remaining pancreatic prosthesis or its removal in the study groups. Secondary endpoints are spontaneous removal of the pancreatic stent, length of hospital stay, rate of follow-up examinations per group, influencing factors, and a possible exploratory analysis.

DETAILED DESCRIPTION:
After study consent, randomization takes place into the standard group (removal of the protective pancreatic stent after 12 hours at the earliest and 10 days at the latest by esophagogastroduodenoscopy/ERCP) or into the intervention group (removal of the protective pancreatic stent after 4 weeks at the earliest, but no later than 3 months).

Both the baseline data and randomization are planned on a secure online platform (http://myresearchmanager.com).

Before removing the pancreatic stent, non-invasive diagnostics may be performed in accordance with hospital standards, and endoscopy may be omitted if the pancreatic stent is found to be displaced.

ELIGIBILITY:
Inclusion Criteria:

* prophylactic pancreatic stent (5Fr 4cm length)
* informed consent

Exclusion Criteria:

* necrotising post-ercp-pancreatitis
* pregnancy/breastfeeding
* Billroth II

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2031-12 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events | From enrollment to the end of treatment at 6 months
  Side effects (number and type) which occur due to the stent insertion, retention after more than 10 days and/or after the removal of the stent

SECONDARY OUTCOMES:
Spontaneous dislocation | From enrollment to the end of treatment 6 months
  Due the examinations by ultrasound and x-ray or endoscopy, the rate of how many patients had a spontaneous dislocation will be evaluated
Follow-up examinations for pancreatic stent detection | From enrollment to the end of treatment at 6 months
  Follow-up examinations for pancreatic stent detection - retention or spontaneous dislocation - by ultrasound, x-ray or endoscopy examination
ERCP procedures | During visit Nr 1 (Day 10 after enrollment)
  Influence of measures taken during ERCP on the probability of spontaneous stent dislocation as well of patients characteristics (pancreaticobiliary disease)
  * questions about procedures made during the ERCP (papillotomy, stent insertion, using metallic stent, balloon dilatation)
  * questions about patients characteristics (chronic pancreatitis, pancreatic tumor, cholangiocarcinoma, stone extraction)
Days of hospital stay | From the date of hospital admission (Day 1) up to hospital discharge, assessed up to 90 days.
  The total number of days participants remain hospitalized from the date of admission until the date of discharge.
Explorative analysis of the collected data | Through study completion, an average of 1 year
  The all data collected will be evaluated and explored for factors influencing our primary endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- Johann Wolfgang Goethe-Universität Frankfurt am Main, Frankfurt, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Michael FA, Feldmann C, Erasmus HP, Kubesch A, Goerguelue E, Knabe M, Abedin N, Heilani M, Hessz D, Graf C, Walter D, Finkelmeier F, Mihm U, Lingwal N, Zeuzem S, Bojunga J, Friedrich-Rust M, Dultz G. A novel ultrasound-based algorithm for the detection of pancreatic stents placed for prophylaxis of post-ERCP pancreatitis: a prospective trial. Ultraschall Med. 2025 Apr;46(2):177-185. doi: 10.1055/a-2407-9651. Epub 2024 Sep 2. PMID 39222928
- [Result] Dultz G, Gerber L, Zeuzem S, Bojunga J, Friedrich-Rust M. Prolonged retention of prophylactic pancreatic stents is not associated with increased complications. Pancreatology. 2019 Jan;19(1):39-43. doi: 10.1016/j.pan.2018.11.011. Epub 2018 Nov 22. PMID 30502123
- [Result] Dumonceau JM, Kapral C, Aabakken L, Papanikolaou IS, Tringali A, Vanbiervliet G, Beyna T, Dinis-Ribeiro M, Hritz I, Mariani A, Paspatis G, Radaelli F, Lakhtakia S, Veitch AM, van Hooft JE. ERCP-related adverse events: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2020 Feb;52(2):127-149. doi: 10.1055/a-1075-4080. Epub 2019 Dec 20. PMID 31863440